CLINICAL TRIAL: NCT01639170
Title: Intra-abdominal Free Air on a Plain Radiograph After Surgery. Could it be a Finding That May Predict Gastrointestinal Perforation?
Brief Title: Abdominal Free Air After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federico II University (Other)
Responsible Party: Principal Investigator, Francesco Milone, Prof. of Surgery. Director of the department, Federico II University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: Federico II-0919
Record Dates: First submitted 2012-07-10; First posted 2012-07-12 (Estimated); Last update posted 2012-07-17 (Estimated); Status verified 2012-06

CONDITIONS: Prediction of Gastrointestinal Perforation
Keywords: Pneumoperitoneum; Free air; Surgery; Perforation; Radiograph
MeSH Terms: conditions — Pneumoperitoneum

ARMS (1):
- subjects undergoing abdominal surgery (Experimental): Subjects who undergone abdominal intervention and reported major symptoms and signs suggestive of gastrointestinal perforation (abdominal pain, leukocytosis, fever) within the third postoperative day.
  Exclusion criteria: inability to consent to the study, age ≤18 yr, certain or probable pregnancy, inability to remain in upright position for more than 10 minutes.
  Interventions: Radiation: chest radiograph

INTERVENTIONS:
Radiation: chest radiograph — All enrolled patients underwent erect chest x-rays assessment. In all cases the diagnosis of pneumoperitoneum was based upon the plain film identification of subdiaphragmatic air on the upright posteroanterior chest radiograph.
  All patients were transported from their hospital rooms to the radiology department in wheelchairs and remained in an upright position for more than 10 min before the chest radiographs were obtained. In all cases upright posteroanterior was obtained with the patient standing, using 183-cm distance, 125 kVp, phototimed exposure, and radiographic film with a wide exposure latitude.
  The disappearance of intraabdominal free gas will be evaluated every 48h and will be defined as the loss of the

SUMMARY:
The aim of this study is to evaluate if the presence of abdominal free air on a plain chest radiograph predicts gastrointestinal perforation. We aimed to enroll all patients undergoing abdominal surgery reporting major symptoms and signs suggestive of gastrointestinal perforation (abdominal pain, leukocytosis, fever) within the third postoperative day.

ELIGIBILITY:
Inclusion Criteria:

* Abdominal surgery and major symptoms and signs suggestive of gastrointestinal perforation within the third postoperative day.

Exclusion Criteria:

* inability to consent to the study, age ≤18 yr, certain or probable pregnancy, inability to remain in upright position for more than 10 minutes.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2011-06; Primary Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
prediction of gastrointestinal perforation | Within 3 days from surgery
  • Prediction of the presence of gastrointestinal perforation by the finding of intra-abdominal free air on a chest radiograph after abdominal surgery

SECONDARY OUTCOMES:
time taken for the absorption of intra-abdominal free air | within 3 days from surgery
  The evaluation of time taken for the absorption of intra-abominal free air and its correlation with age, sex, body mass index, previous surgery, operative time, type of surgery and use of peritoneal drainage tubes.
  The disappearance of intra-abdominal free gas was defined as the loss of the gas bubble under the domes of the hemidiaphragms on an erect chest radiograph

CONTACTS AND LOCATIONS:
Locations (1):
- "Federico II" University, Naples, Italy, Italy

REFERENCES:
- [Result] Tang CL, Yeong KY, Nyam DC, Eu KW, Ho YH, Leong AF, Tsang CB, Seow-Choen F. Postoperative intra-abdominal free gas after open colorectal resection. Dis Colon Rectum. 2000 Aug;43(8):1116-20. doi: 10.1007/BF02236559. PMID 10950010
- [Result] Hope WW, Heniford BT, Norton HJ, Lincourt AE, Teigland CM, Kercher KW. Duration and clinical significance of radiographically detected "free air" after laparoscopic nephrectomy. Surg Laparosc Endosc Percutan Tech. 2009 Oct;19(5):415-8. doi: 10.1097/SLE.0b013e3181b6bff3. PMID 19851274
- [Result] BRYANT LR, WIOT JF, KLOECKER RJ. A STUDY OF THE FACTORS AFFECTING THE INCIDENCE AND DURATION OF POSTOPERATIVE PNEUMOPERITONEUM. Surg Gynecol Obstet. 1963 Aug;117:145-50. No abstract available. PMID 14048004
- [Result] Nielsen KT, Lund L, Larsen LP, Knudsen P. Duration of postoperative pneumoperitoneum. Eur J Surg. 1997 Jul;163(7):501-3. PMID 9248983
- [Result] Gayer G, Jonas T, Apter S, Amitai M, Shabtai M, Hertz M. Postoperative pneumoperitoneum as detected by CT: prevalence, duration, and relevant factors affecting its possible significance. Abdom Imaging. 2000 May-Jun;25(3):301-5. doi: 10.1007/s002610000036. PMID 10823456
- [Result] Schauer PR, Page CP, Ghiatas AA, Miller JE, Schwesinger WH, Sirinek KR. Incidence and significance of subdiaphragmatic air following laparoscopic cholecystectomy. Am Surg. 1997 Feb;63(2):132-6. PMID 9012426
- [Result] Millitz K, Moote DJ, Sparrow RK, Girotti MJ, Holliday RL, McLarty TD. Pneumoperitoneum after laparoscopic cholecystectomy: frequency and duration as seen on upright chest radiographs. AJR Am J Roentgenol. 1994 Oct;163(4):837-9. doi: 10.2214/ajr.163.4.8092019.
- [Result] Earls JP, Dachman AH, Colon E, Garrett MG, Molloy M. Prevalence and duration of postoperative pneumoperitoneum: sensitivity of CT vs left lateral decubitus radiography. AJR Am J Roentgenol. 1993 Oct;161(4):781-5. doi: 10.2214/ajr.161.4.8372757.
- [Derived] Milone M, Di Minno MN, Bifulco G, Maietta P, Sosa Fernandez LM, Musella M, Iaccarino V, Buccelli C, Nappi C, Milone F. Diagnostic value of abdominal free air detection on a plain chest radiograph in the early postoperative period: a prospective study in 648 consecutive patients who have undergone abdominal surgery. J Gastrointest Surg. 2013 Sep;17(9):1673-82. doi: 10.1007/s11605-013-2282-6. Epub 2013 Jul 20. PMID 23877326